CLINICAL TRIAL: NCT06594666
Title: Clinical Study on the Effectiveness and Safety of Visual Training for Improving Intermittent Exotropia Visual Function
Brief Title: Visual Training for Improving Intermittent Exotropia Visual Function
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: QX-2024-A-012
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Intermittent Exotropia; Visual Functions
Keywords: visual training; visual function; intermittent exotropia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VR/AR visual training group (Experimental): Wear glasses for correction combined with VR/AR visual training in the first 6 months, and terminate the training for follow-up observation in the last 6 months. Regular follow-up every 3 months, with a total follow-up time of 1 year.
  Interventions: Device: VR/AR visual training group
- control group (No Intervention): No intervention, simply wearing glasses for correction, followed up every 3 months for a total of 12 months.

INTERVENTIONS:
Device: VR/AR visual training group — Wear glasses for correction combined with VR/AR visual training in the first 6 months, and terminate the training for follow-up observation in the last 6 months. Regular follow-up every 3 months, with a total follow-up time of 1 year.
  Arms: VR/AR visual training group

SUMMARY:
The goal of this clinical tral is to investigate that if VR/AR visual training can improve the visual function in children with intermittent exotropia.

The main question it aims to answer is :

Does the VR/AR visual training can enhance stereoscopic vision function in children with intermittent exotropia.

Researchers will compare intervention group to control group to see if VR/AR visual training could enhance stereoscopic vision function in children with intermittent exotropia.

Participants will:

The intervention group will receive 20 minutes of VR/AR visual training once a day for a period of one year.

Follow up check ups at the hospital every 3 months. Keep a diary of the values of stereoscopic vision function and Newcastle Control Score.

ELIGIBILITY:
Inclusion Criteria:

Aged 6 to 14 years. Intermittent exotropia meeting all of the following criteria: Exodeviation at least 10Δ at distance measured by the prism and alternate cover test, near deviation does not exceed distance deviation by more than 10Δby prism and alternate cover test, mean distance Newcastle Control Score (NCS)≥2 points (mean of 3 assessments during the examination).

Refractive error between -5.00 D < spherical equivalents (SEs) ≤ -1.00 D, astigmatism ≤1.50D, anisometropia ≤1.5D, best visual acuity in each eye of 1.0.

Not receiving any other form of strabismus or myopia treatment within 3 months. Willing to follow the research plan and participate in the entire research process.

Participants and guardians agree to be randomly assigned and sign an informed consent form.

Exclusion Criteria:

Vertical strabismus; Diagnosed with other eye diseases or visual abnormalities such as strabismus, amblyopia, etc; Existence of cognitive or learning disabilities that may affect the effectiveness of training; patients with neurological disorders; Unable to cooperate with eye examination and follow-up work.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 78 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
changes in stereoscopic vision function after 6 month | 6 months after baseline
  Compare whether the intervention group has better stereoscopic vision function than the control group after 6 months
changes in stereoscopic vision function after 12 month | 12 month after baseline
  Stop the intervention group training after 6 months and observe for another 6 months to see if there will be a decrease in stereoscopic vision function.